CLINICAL TRIAL: NCT02205788
Title: Feasibility of Biodynamic Imaging for Predicting Effect of Gemcitabine and Nab-paclitaxel on Metastatic Adenocarcinoma of the Pancreas
Brief Title: Feasibility of Biodynamic Imaging for Predicting Therapeutic Effect in Metastatic Adenocarcinoma of the Pancreas
Status: Withdrawn | Type: Observational
Sponsor: Patrick Joseph Loehrer Sr. (Other)
Responsible Party: Sponsor-Investigator, Patrick Joseph Loehrer Sr., Professor, Indiana University
Organization: Indiana University (Other)
Other Study IDs: IUCRO-0479; 1405049285 (Other: Indiana University IRB)
Record Dates: First submitted 2014-07-10; First posted 2014-07-31 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — core needle biopsy of tumor
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if you can use an assay on tumor samples to see different patterns in response to the same chemotherapy treatment.

DETAILED DESCRIPTION:
To examine the feasibility of using biodynamic imaging (BDI) as a chemosensitivity assay on fresh tumor samples obtained by core needle biopsy from patients planned to receive routine care gemcitabine and nab-paclitaxel for treatment of metastatic adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an informed consent and authorization for release of health information for research
2. ≥ 18 years old at time of consent
3. Patients with a diagnosis of metastatic pancreatic cancer (mPC) who have not received prior combination chemotherapy. Exception: prior adjuvant chemoradiation with fluorouracil or gemcitabine is allowed.
4. Patients considered for routine care treatment with gemcitabine and nab-paclitaxel (allowed to receive other experimental therapy with gem/nab backbone if participating in another clinical trial)
5. Measurable disease by RECIST v1.1 criteria
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
7. Willingness to undergo transcutaneous core needle biopsy of metastatic tumor for research purposes
8. Women are eligible to participate if they are of non-childbearing potential or have documentation of a negative pregnancy test (serum or urine β-hCG) within 1 week of the start of protocol treatment.
9. Women and men of childbearing potential must agree to use adequate, highly effective contraceptive measures during protocol treatment
10. Laboratory values: Platelets ≥ 100 K/mm3 international normalized ratio (INR) < 1.2, Partial thromboplastin time (PTT) in normal range, Cr < 2.0, Total bilirubin < 2 times upper limit normal (ULN), transaminases < 5 times ULN

Exclusion Criteria:

1. History of abnormal bleeding with minor procedures or documented platelet aggregation disorder such as VonWillebrand disease
2. Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic and Cancer Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
BDI as a chemosensitivity assay on fresh tumor samples | up to 336 days
  To examine the feasibility of using BDI as a chemosensitivity assay on fresh tumor samples obtained by core needle biopsy from patients planned to receive routine care gemcitabine and nab-paclitaxel for treatment of metastatic adenocarcinoma of the pancreas.

SECONDARY OUTCOMES:
BDI patterns and results with Response Evaluation Criteria | up to 336 days
  To compare BDI patterns consistent with chemotherapy response ex-vivo to response to chemotherapy as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bert O'Neil, MD, Principal Investigator — Indiana University